CLINICAL TRIAL: NCT05923177
Title: SPECT Imaging of Human Epidermal Growth Factor Receptor 2 (HER2) Expression in Breast Cancer Using Iodine -123-labelled Designed Ankyrin Repeat Proteins HE3-G3 ([123I] I-(HE)3-G3)
Brief Title: Molecular Imaging of HER2 Expression in Breast Cancer Using [123I] I-(HE)3-G3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: [123I] I-(HE)3-G3
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Primary Breast Cancer
MeSH Terms: interventions — Iodine-123

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The tested injected doses of [123I] I-(HE)3-G3 3000 μg (Experimental): At least five (5) evaluable subjects with HER2-positive status and at least five (5) subjects with HER2-negative status have to be enrolled in the study for each tested protein dose. The tested injected dose 3000 μg.
  Subjects withdrawn from the study for any reason will be replaced
  Interventions: Drug: SPECT

INTERVENTIONS:
Drug: SPECT — One single injection of [123I] I-(HE)3-G3, followed by gamma camera imaging directly postinjection and after 2, 4, 6, 24 and 48 hours.
  Other Names: [123I] I-(HE)3-G3

SUMMARY:
The study should evaluate distribution of [123I] I-(HE)3-G3 in patients with primary HER2-positive and HER2-negative breast cancer

DETAILED DESCRIPTION:
Overall goal of the project: To determine HER2 expression level in primary breast cancer before neoadjuvant system therapy.

Phase I. Distribution of HE3-G3 ([123I] I-(HE)3-G3) in patients with primary breast cancer. The study should evaluate distribution of HE3-G3 ([123I] I-(HE)3-G3) in patients with primary HER2-positive and HER2-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 years of age
2. Availability of results from HER2 status previously determined on material from the primary tumor and metastatic LN, either a. HER2-positive, defined as a DAKO HercepTest™ score of 3+ or FISH positive or b. HER2-negative, defined as a DAKO HercepTest™ score of 0 or 1+; or else if 2+ then FISH negative
3. Hematological, liver and renal function test results within the following limits:

   * White blood cell count: > 2.0 x 109/L
   * Hemoglobin: > 80 g/L
   * Platelets: > 50.0 x 109/L
   * ALT, ALP, AST: =< 5.0 times Upper Limit of Normal
   * Bilirubin =< 2.0 times Upper Limit of Normal
   * Serum creatinine: Within Normal Limits
4. A negative pregnancy test for all patients of childbearing potential. Sexually active women of childbearing potential participating in the study must use a medically acceptable form of contraception for at least 30 days after study termination
5. Subject is capable to undergo the diagnostic investigations to be performed in the study
6. Informed consent

Exclusion Criteria:

1. Any system therapy (chemo-/targeted therapy)
2. Second, non-breast malignancy
3. Active current autoimmune disease or history of autoimmune disease
4. Active infection or history of severe infection within the previous 3 months (if clinically relevant at screening) 4. Known HIV positive or chronically active hepatitis B or C
5. Administration of other investigational medicinal product within 30 days of screening
6. Ongoing toxicity > grade 2 from previous standard or investigational therapies, according to US National Cancer Institute's

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with primary breast cancer
Enrollment: 10 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Gamma camera-based whole-body [123I] I-(HE)3-G3 uptake value (%) | 6 hours
  Whole-body [123I] I-(HE)3-G3 uptake coinciding with normal organs and tissues will be assessed using gamma camera and calculated as percentage (%) of the injected dose of the radiopharmaceutical
SPECT-based [99mTc]Tc-G3-(G3S)3C uptake value in tumor lesions (counts) [123I] I-(HE)3-G3 uptake coinciding with tumor lesions will be assessed using single-photon emission computed tomography and measured in counts | 6 hours
  SPECT-based [99mTc]Tc-G3-(G3S)3C uptake value in tumor lesions (counts) [123I] I-(HE)3-G3 uptake coinciding with tumor lesions will be assessed using single-photon emission computed tomography and measured in counts
SPECT-based [123I] I-(HE)3-G3 background uptake value (counts) | 6 hours
  Focal uptake of [123I] I-(HE)3-G3 in the regions without pathological findings will be assessed with SPECT and measured in counts
Tumor-to-background ratio (SPECT) | 6 hours
  The SPECT-based tumor-to-background ratio will be calculated as follows: the value of [123I] I-(HE)3-G3 uptake coinciding with tumor lesions (counts) will be divided by the value of [123I] I-(HE)3-G3 uptake coinciding with the regions without pathological findings (counts)

SECONDARY OUTCOMES:
Safety attributable to [123I] I-(HE)3-G3 injections (physical examination) (% of cases with abnormal findings relative to baseline) | 48 hours
  The safety attributable to [123I] I-(HE)3-G3 injections will be evaluated based on the assessments of physical examination (% of cases with abnormal findings relative to baseline)
Safety attributable to [123I] I-(HE)3-G3 injections (vital signs) (% of cases with abnormal findings relative to baseline) | 48 hours
  The safety attributable to [123I] I-(HE)3-G3 injections will be evaluated based on the assessments of vital signs (% of cases with abnormal findings relative to baseline)
Safety attributable to [123I] I-(HE)3-G3 injections (ECG) (% of cases with abnormal findings relative to baseline) | 48 hours
  The safety attributable to [123I] I-(HE)3-G3 injections will be evaluated based on the assessments of ECG (% of cases with abnormal findings relative to baseline)
Safety attributable to [123I] I-(HE)3-G3 injections (laboratory tests) (% of cases with abnormal findings relative to baseline) | 48 hours
  The safety attributable to [123I] I-(HE)3-G3 injections will be evaluated based on the blood and urine laboratory tests (% of cases with abnormal findings relative to baseline)
Safety attributable to [123I] I-(HE)3-G3 injections (% of incidence and severity of adverse events) | 48 hours
  The safety attributable to [123I] I-(HE)3-G3 injections will be evaluated based on the rate of adverse events (%)

CONTACTS AND LOCATIONS:
Overall Officials: Olga Bragina, Dsc, Principal Investigator — Tomsk NRMC
Locations (1):
- TomskNRMC, Tomsk, Russia